CLINICAL TRIAL: NCT00780260
Title: Case Management Alternatives for African American Women at High Risk for HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R01DA013131-06A2 (NIH); R01DA013131-06A2 (NIH)
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: HIV
Keywords: HIV/AIDS; African Americans; Women; Case Management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 5 session strengths-based case management intervention delivered by a professional case manager and a peer support specialist team
  Interventions: Behavioral: strengths-based case management
- 2 (Active Comparator): 5 session strengths-based case management intervention delivered by a professional case manager.
  Interventions: Behavioral: strengths-based case management

INTERVENTIONS:
Behavioral: strengths-based case management — 5 session individual strengths-based case management; peer-involvement v. no peer involvement

SUMMARY:
The purpose of this study is to test two innovative case management approaches designed to increase linkages and engagement with drug abuse treatment, HIV-related care, and other health services among an underserved population of African American women at risk for HIV.

DETAILED DESCRIPTION:
The study is fundamentally concerned with the implementation and evaluation of theoretically-based, culturally appropriate case management interventions targeting individual, social and environmental factors among highly vulnerable African American women. The research is designed to test innovative, comprehensive approaches to HIV prevention/intervention through case management driven service linkage and engagement. Testing new approaches to intervention with African-American women at high risk for HIV addresses a particularly urgent public health need in Miami, as well as other large metropolitan areas, where officials continue to document epidemic rates of HIV/AIDS clustered in urban, impoverished African-American communities.

Comparison: Participants will be randomly assigned to: a Strengths-Based / Professional Only Condition in which clients participate in a "strengths-based" case management approach; or, a Strengths-Based / Professional/Peer Condition in which a team composed of: a) a credentialed, professional case manager and b) a recovering addict peer - both trained in "strengths-based" case management techniques - develop and facilitate the implementation of a service plan.

ELIGIBILITY:
Inclusion Criteria:

* Current substance abuse
* Current high-risk sexual behavior
* African American racial identification

Exclusion Criteria:

* Non resident of Miami-Dade county

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 562 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Substance abuse treatment linkage at 3 months | 3 months
Substance abuse treatment engagement at 6 months | 6 months
HIV related care at 3 and 6 months | 3 and 6 months
Other health service utilization at 3 and 6 months | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hilary L Surratt, Ph.D., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Miami, Florida, United States